Effect of Monazite Sands in Patients with Osteoarthritis of the Knee

Ethical committee Protocol No: 3.160.891

Withdrawal\_log

Documente date: May 3<sup>rd</sup>, 2019

## SUBJECT WITHDRAWAL/TERMINATION LOG

**Study brief Title:** Effects of Sand Treatment on Osteoarthritis

Official Title: Effect of Monazite Sands in Patients With Osteoarthritis of the Knee

Ethical committee Protocol No: 3.160.891 Unique Protocol ID: T015-M02-2019AF002

| S.No | Subject ID | Date of withdrawal/<br>termination<br>(dd/mm/yyyy) | Reason for withdrawal/<br>termination <sup>1</sup> | Notified date<br>(dd/mm/yyyy) | Investigator<br>Initials and Date | Comments |
|---|---|---|---|---|---|---|

Legend: 1. Reasons for removal of patients from the study: (A) Underwent knee surgery during the course of the research; (B) Subjected to joint infiltration with corticoids or any other type of intra-articular medication; (C) Failure to attend more than 3 consecutive exposures; (D) Intolerance to heat or any type of discomfort during exposure to sand.

| Signature of the Principal Investigator: | Date: |
|------------------------------------------|-------|